CLINICAL TRIAL: NCT05787795
Title: Identifying and Characterizing Preclinical MS
Acronym: DREAM
Status: Recruiting | Type: Observational
Sponsor: Yale University (Other)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Other Study IDs: 2000032952
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood and gingival swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: biological samples — blood draw, oral swab, optional stool samples, spinal fluid sample, fat biopsy, tonsil biopsy, lymph node tissue sample, MRI

SUMMARY:
The purpose of this research study is to try and identify risk factors and biologic changes that suggest that someone may go on to develop multiple sclerosis before a person has shown any symptoms of the disease.

DETAILED DESCRIPTION:
The purpose of this study is to try and learn how to identify multiple sclerosis (MS) before it causes any neurologic symptoms. By the time MS causes symptoms, the disease has often been causing damage under the surface for years. Because early treatment of MS helps prevent long term disability from the disease, the investigators are hypothesizing that if MS could be detected (and treated) before symptoms start, the disease might be preventable.

The investigators believe that people who go on to develop MS have changes in their immune systems long before they have symptoms. Some of these changes might be in "hidden" parts of the body, like lymph nodes or fat tissue. The investigators want to study people who have risk factors for MS to try and learn to detect very early signs of disease.

Study procedures will include:

All study participants will undergo a blood draw and an oral swab; they will also complete baseline questionnaires All study participants will be contacted approximately once per year and asked to complete some additional questionnaires All study participants may be asked to donate repeat blood/oral swab specimens or stool specimens over time on an ad hoc basis Study participants who agree will undergo additional optional procedures to study the immune system in different parts of the body.

The optional procedures include:

Lumbar punctures (to obtain spinal fluid) Tonsil biopsy Fat biopsy (to obtain fat cells) Lymph node biopsy (to obtain lymph node tissues with immune cells) Traditional brain MRI Low-field (portable) brain MRI

One in-person visit is required. There will also be annual phone/email contact, which may take up to 30 minutes The required in-person visit will take approximately 1 hour total. Anyone who agrees to donate follow up biospecimens, undergo a procedure, or undergo an MRI will have additional in-person visits Optional visits for donating biospecimens, having a procedure or getting an MRI may take longer (up to 3 hours), depending on what is happening during the visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Having one or more risk factors for multiple sclerosis, including one or more of the below:

  * Individuals known to have a radiologically isolated syndrome
  * Individuals with a family history of multiple sclerosis (first degree family member)
  * Individuals with personal risk factors, which are known to include smoking, obesity, Epstein Barr virus infections, Vitamin D deficiency, genetic risk score

Exclusion Criteria:

* Currently pregnant
* Diagnosis of multiple sclerosis or any ongoing, systemic autoimmune disease
* Ongoing treatment with immunosuppressive medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with risk factors for MS (based on personal demographics, past medical history, or family history) will be recruited to provide clinical information and biospecimens serially over time.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2032-06-30 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
To build a machine learning model of risk prediction | ongoing prospective study
  to build a risk prediction model that estimates future risk of MS built using large datasets of biologic and clinical data collected during the study.

SECONDARY OUTCOMES:
Individual data types collected | ongoing prospective study
  Microbiome data, immune phenotyping and functional analysis for blood, CSF, adipose tissue, measurement of other known and developing biomarkers of MS, patient reported health outcomes will be compiled to potentially identify early, systemic changes that are associated with a future risk of multiple sclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Longbrake, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, North Haven, Connecticut, United States